CLINICAL TRIAL: NCT05362890
Title: The Role of the Device Operating Under the Continuous Positive Airway Pressure in the Recovery Process of Cochlear Receptor Cells in Patients With Obstructive Sleep Apnea
Brief Title: The Role of the Device Operating Under the Continuous Positive Airway Pressure in the Recovery Process of Cochlea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mirjana Grebenar Cerkez (Other)
Responsible Party: Sponsor-Investigator, Mirjana Grebenar Cerkez, Mirjana Grebenar Cerkez, M.D. ENT specialist, audiologist, Osijek University Hospital
Organization: Osijek University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OSIJEKUH-OAE-101
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Cochlear receptor cells; Hearing; CPAP device; Hypoxia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with obstructive sleep apnea (Experimental): Patients with OSAS who have been previously examined by a neurologist for sleep disorders, have undergone polysomnography, and have been diagnosed with moderate severe obstructive sleep apnea according to the AHI index
  Interventions: Device: DEVICE OPERATING UNDER THE CONTINOUS POSITIVE AIRWAY PRESSURE
- Control Group (No Intervention): The control group will consist of subjects in whom specific questionnaires excluded the existence of obstructive sleep apnea.

INTERVENTIONS:
Device: DEVICE OPERATING UNDER THE CONTINOUS POSITIVE AIRWAY PRESSURE — The principle of operation is to prevent the closure and the narrowing of the structures of the upper respiratory tract by applying positive pressure. The device consists of a mask that protects the nose and/or mouth, a tube that connects the mask to the monitor and a monitor that blows air into the tube. A pressure in the range of 4 to 20 cm water is applied, depending on the individual needs of the patient to keep the airway open. The use is considered to be effective when the patient uses it continuously for at least 4 hours at bedtime. Today's modern devices have memory cards for storing data on the regularity and time of use of the device during the night and the efficiency of the device itself. For therapy to be considered effective, the number of apneas and hypopneas must be less than 5 per hour of sleep.
  Other Names: CPAP
  Arms: Patients with obstructive sleep apnea

SUMMARY:
Hypothesis: Patients with obstructive sleep apnea syndrome (OSAS) have cochlear receptor cells damage because of prolonged, recurrent hypoxia. The use of devices operating under the continous positive airway pressure (CPAP) leads to the recovery of cochlear receptor cells.

Aims:

1. To determinate whether there is cochlear receptor cells damage in OSAS patients depending on the degree of the disease
2. Investigate whether the use of ventilation devices with continuous positive pressure and constant oxygen pressure in the airways can lead to the recovery of the cochlear receptor cells Participants and Methods: The investigation work will be designed as original scientific research- prospective cohort study at Department od Otorhinolaryngology and Head and Neck Surgery, University Hospital Center Osijek.

The participants will be divided in two groups: target group with obstructive sleep apnea (n45) and control group with healthy individuals (n32).

Research plan: All participating in this study will complete the following questionnaires: STOP- BANG and Epworth drowsiness scale. Subjects of the target group with moderate or severe obstructive sleep apnea will be referred to an otorhinolaryngologist audiologist for complete examination and processing after examination by a neurologist. These participants will be examined by an audiologist after 6-8 months of continuous and adequate use of the CPAP device for reevaluation. Participants of a control group will be patients examined or treated in Department of Otorhinolaryngology and Head and Neck surgery for other diseases in whom specific questionnaires excluded the existence of obstructive sleep apnea. Audiological diagnostics will be performed on all patients on the same devices of the Department of Audiology and Phoniatrics .

Expected scientific contribution: To prove the existence of receptor hearing impairment in the patients with obstructive sleep apnea; and then to prove that the use of a of continuous positive airway pressure with constant oxygen pressure in patients with OSAS using CPAP devices leads to the recovery of the cochlear receptor cells whose damage occurred as a result prolonged recurrent hypoxia. In addition, to determine the importance of a broader diagnostic processing of patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
The participants will be divided in two groups: target (n45) and control group (n32). The target group will consist of patients with OSAS who have been previously examined by a neurologist for sleep disorders, have undergone polysomnography, and have been diagnosed with moderate or severe obstructive sleep apnea according to the Apnea Hypopnea Index (AHI) : the number of apneas or hypopneas recorded during the study per hour of sleep. It is generally expressed as the number of events per hour./hypopnea index). The control group will consist of subjects in whom specific questionnaires excluded the existence of obstructive sleep apnea. Exclusive criteria are age less than 18 years, persons with previous neurootological diseases that required surgical treatment, and persons who deviate from the research protocol.

Research plan: All participants in this study will complete the following questionnaires:

1. STOP-BANG :

   Snoring ? Do you Snore Loudly (loud enough to be heard through closed doors or your bed-partner elbows you for snoring at night)? Yes or No Tired ? Do you often feel Tired, Fatigued, or Sleepy during the daytime (such as falling asleep during driving or talking to someone)? Yes or No Observed ?Has anyone Observed you Stop Breathing or Choking/Gasping during your sleep ? Yes or No Pressure ? Do you have or are being treated for High Blood Pressure ? Yes or No Body Mass Index more than 35 kg/m2? Yes or No Age older than 50 ? Yes or No Neck size large ? (Measured around Adams apple) Is your shirt collar 16 inches / 40cm or larger? Yes or No Gender = Male ? Yes or No Results: OSA - Low Risk : Yes to 0 - 2 questions OSA - Intermediate Risk : Yes to 3 - 4 questions OSA - High Risk : Yes to 5 - 8 questions or Yes to 2 or more of 4 STOP questions + male gender or Yes to 2 or more of 4 STOP questions + BMI > 35kg/m2 or Yes to 2 or more of 4 STOP questions + neck circumference 16 inches / 40cm
2. Epworth sleepiness scale How Sleepy Are You?

How likely are you to doze off or fall asleep in the following situations? You should rate your chances of dozing off, not just feeling tired. Even if you have not done some of these things recently try to determine how they would have affected you. For each situation, decide whether or not you would have:

* No chance of dozing =0
* Slight chance of dozing =1
* Moderate chance of dozing =2
* High chance of dozing =3

Write down the number corresponding to your choice:

Sitting and reading · Watching television · Sitting inactive in a public place (e.g., a theater ora meeting) As a passenger in a car for an hour without a break Lying down to rest in the afternoon when circumstances permit Sitting and talking to someone · Sitting quietly after a lunch without alcohol · In a car, while stopped for a few minutes in traffic

Interpretation:

0-7:It is unlikely that you are abnormally sleepy. 8-9:You have an average amount of daytime sleepiness. 10-15:You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention. 16-24:You are excessively sleepy and should consider seeking medical attention.

Subjects of the target group with severe obstructive sleep apnea will be referred to an otorhinolaryngologist audiologist for complete neurootological examination and processing after an examination by a neurologist. These participants will be examined by an audiologist after 6-8 months of continuous and adequate use of the CPAP device for reevaluation. Participants of a control group will be patients examined or treated in Department of Otorhinolaryngology and Head and neck surgery for other diseases in whom specific questionnaires (STOP BANG and Epworth sleepiness scale excluded the existence of obstructive sleep apnea. Audiological diagnostics will be performed on all patients on the same devices of the Department of Audiology and Phoniatrics and it will include:

* A Puretone audiometry (subjective method of hearing testing using a device called an audiometer; the test is performed at frequencies from 125 to 8000 Hz, where earphones are placed on the ear for air conduction and vibration on the mastoid which records bone conduction; the sound is emitted from quieter to louder, the lowest value the respondent hears is considered the hearing threshold);
* A tympanometry (a method of testing the pressure of the middle ear that is performed by placing a three-channel probe, speaker, microphone and pressure-changing channel in the subject's external ear canal; the method is objective, but the movement and the swallowing can affect the result; the test result is a curve which shows how much sound released into the external ear canal bounced off the eardrum and returned to the microphone);
* An Acoustic Stapedius Reflex (diagnostic method that can be performed without the cooperation of the subject; the principle of the method is based on the fact that when a sound of a certain intensity is released into the ear, the muscle in the middle ear is reflexively compressed and the flexibility of auditory bones in the middle ear changes in order to reduce the conduction of sound to the inner ear, which serves as a protective reflex from excessive noise; in the case of a receptor hearing damage, the volume required to trigger the reflex is lower than usual);
* An Auditory Brainstem Response (neurootological method for examining the response of the VIII cerebral nerve and auditory pathway in the brainstem to acoustic stimulation, i.e. audiometry using evoked brainstem responses; it is performed using a headset which gives a large number of short <1 ms click stimuli, at a speed of 20/s, a total of 2000 stimuli, the electrical activity of the VIII nerve and auditory structures in the brainstem is registered, which occurs in the interval of 1.5-10 ms after a repeated stimulus of a certain intensity);
* An Otoacoustic Emission (TEOAE and DPOAE) is an objective method; it is performed by placing a probe with a plastic insertion into the subject's external ear canal and by recording the returning sound (an echo) with a sensitive microphone; the echo occurs in cases where the middle ear and cochlea i.e. cochlear receptor cells are healthy; the TEOAE shows the status of the whole cochlea, while the DPOAE examines more specific frequency regions).

ELIGIBILITY:
Inclusion Criteria:

* Patients with OSAS who have been previously examined by a neurologist for sleep disorders, have undergone polysomnography, and have been diagnosed with moderate or severe obstructive sleep apnea according to the AHI index
* Healthy individuals for control group that will consist of subjects in whom specific questionnaires excluded the existence of obstructive sleep apnea.

Exclusion Criteria:

* age less than 18 years,
* persons with previous neurootological diseases that required surgical treatment
* persons who deviate from the research protocol.

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Hearing test Otoacoustic Emission (TEOAE and DPOAE) | 45 minutes for each participant initialy and then after six to eight months of using device new measurement
  Objective analysis of hearing using otoacoustic emission in decibels. It is an objective method; it is performed by placing a probe with a plastic insertion into the subject's external ear canal and by recording the returning sound (an echo) with a sensitive microphone; the echo occurs in cases where the middle ear and cochlea i.e. cochlear receptor cells are healthy; the TEOAE shows the status of the whole cochlea, while the DPOAE examines more specific frequency regions.

CONTACTS AND LOCATIONS:
Overall Officials: Darija Birtic, Study Chair — Department of Otorhinolaryngology and Head and Neck Surgery Osijek
Locations (1):
- Department of Otorhinolaryngology and Head and Neck Surgery, University Hospital Center Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Plan is to share the results of pure tone audiometry and results of otoacoustic emission for each individuals in the study
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be available upon completion of research for 12 months long
Access Criteria: The information will be shared with other potential researchers for further analyses